CLINICAL TRIAL: NCT04143724
Title: A Phase 2a Study to Evaluate the Safety and Pharmacokinetics of Luspatercept (ACE-536) in Pediatric Participants With Beta (β)-Thalassemia
Brief Title: Study of Safety & PK of Luspatercept (ACE-536) in Pediatric Participants With Beta (β)-Thalassemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-B-THAL-004; U1111-1241-4168 (Other: WHO); 2022-502499-22 (Other: EU CT Number)
Record Dates: First submitted 2019-10-02; First posted 2019-10-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Beta-Thalassemia
Keywords: ACE-536; Luspatercept; Pharmacokinetics; Beta-Thalassemia; Red Blood Cell Transfusion
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: TD Dose Escalation Cohort: 12 to < 18 years Luspatercept 0.75 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 2: TD Dose Escalation Cohort: 12 to < 18 years: Luspatercept 1.0 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 3: TD Dose Expansion Cohort: 12 to <18 years Luspatercept 1.0 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 4: TD Dose Escalation Cohort: 6 to < 12 years Luspatercept 1.0 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 5: TD Dose Escalation Cohort: 6 to <12 years Luspatercept 1.2 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 6: NTD Dose Confirmation Cohort: 12 to < 18 years Luspatercept 1.0 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 7: NTD Dose Expansion Cohort: NTD 12 to < 18 years (Experimental)
  Interventions: Drug: ACE-536
- Cohort 8: NTD Dose Escalation Cohort: 6 to < 12 years Luspatercept 1.0 mg/kg (Experimental)
  Interventions: Drug: ACE-536
- Cohort 9: NTD Dose Escalation Cohort: 6 to < 12 years Luspatercept 1.2 mg/kg (Experimental)
  Interventions: Drug: ACE-536

INTERVENTIONS:
Drug: ACE-536 — Specified dose on specified days
  Other Names: Luspatercept; BMS-986346

SUMMARY:
This is a Phase 2a study to evaluate the safety and pharmacokinetics (PK) of luspatercept in pediatric participants with β-thalassemia.

The study will be conducted in 2 parts for both transfusion-dependent (TD) and non-transfusion-dependent (NTD) β-thalassemia participants: TD Part A will be in adolescent participants aged 12 to <18 years with two dose escalation cohorts, followed by a dose expansion cohorts. NTD Part A will be conducted in the same age group participants as TD Part A with dose confirmation and expansion cohorts. After Part A TD participants have completed at least one year of treatment, all available safety data from Part A adolescent participants will be evaluated before initiating TD and NTD Part B in the age group from 6 to <12 years old. Part B will consist of two dose escalation cohorts for TD and two dose escalation cohorts for NTD.

Upon completion of the Treatment Period, participants of any cohort who are benefiting from the study treatment, will be offered the opportunity to continue luspatercept treatment in the Long-term Treatment Period for up to 5 years from their first dose.

Participants who discontinue study treatment at any time will continue in the Posttreatment Follow-up Period for at least 5 years from their first dose of luspatercept, or 3 years from their last dose, whichever occurs later, or until they withdraw consent/assent, are lost to follow-up, or the End of Trial, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Participants must be 6 years to < 18 years of age at the time of signing the informed consent form (ICF)/informed assent form (IAF).
* Participants (and when applicable, parent/legal representative) must understand and voluntarily sign an ICF/IAF prior to conducting any study-related assessments/procedures.
* Participants (and when applicable, parent/legal representative) is willing and able to adhere to the study visit schedule and other protocol requirements.
* Participants must have documented diagnosis of β-thalassemia or Hemoglobin E/β-thalassemia.
* Transfusion dependence (TD):

  a. TD participant i. Participant is regularly transfused, defined as: ≥ 4 RBC transfusion events in the 24 weeks prior to enrollment with no transfusion-free period ≥ 42 days during that period.

Note: For the purpose of the study, transfusions administered over 2 or 3 consecutive days are considered as part of a single transfusion event. Participant must have a history of regular transfusions for at least 2 years.

b. NTD participant (ex-US sites only) i. Participant must have received < 4 RBC transfusion events in the 24 weeks prior to enrollment.

ii. Participant must not be on a regular transfusion program and must be RBC transfusion-free for at least 8 weeks prior to enrollment.

iii. Participant must have mean baseline hemoglobin ≤ 10 g/dL, based on a minimum of 2 measurements ≥ 1 week apart within 4 weeks prior to enrollment; hemoglobin values within 21 days post- transfusion will be excluded.

* Participants have Karnofsky (age ≥16 years) or Lansky (age < 16 years) performance status score ≥ 50 at screening.
* Female children of childbearing potential (FCCBP), individuals of childbearing potential (IOCBP), and male (as assigned at birth) participants that have reached puberty (and when applicable, parent/legal representative) must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction.
* Female children of childbearing potential, defined as females who have achieved menarche and/or breast development in Tanner Stage 2 or greater and have not undergone a hysterectomy or bilateral oophorectomy and individuals of childbearing potential (IOCBP) defined as a sexually mature woman who has achieved menarche at some point, has not undergone a hysterectomy or bilateral oophorectomy and has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) must meet the following conditions below (Note: Secondary amenorrhea from any cause does not rule out childbearing potential):
* Medically supervised serum pregnancy tests with a sensitivity of at least 25 mIU/mL must be conducted in Female children of childbearing potential (FCCBP)/ individuals of childbearing potential (IOCBP), including those who commit to complete abstinence. Female children of childbearing potential/ individuals of childbearing potential (IOCBP) must have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy (one of these tests should be performed by central laboratory). Female children of childbearing potential/ individuals of childbearing potential (IOCBP) must agree to ongoing pregnancy testing during the course of the study at the End of Treatment (EOT) visit and at the 9-week Safety Follow-up visit.
* Female participants must, as appropriate to age and at the discretion of the site Investigator, either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective** contraception without interruption, 28 days prior to starting IP, during the study therapy (including dose interruptions), and for 12 weeks (approximately 5 times the mean terminal t1/2 of luspatercept based on multiple-dose PK data) after discontinuation of study therapy.
* Male (as assigned at birth) participants, as appropriate to age and the discretion of the study physician:

  * Must practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a synthetic or latex condom during sexual contact with a pregnant female or a Female children of childbearing potential (FCCBP)/ IOCBP while participating in the study, during dose interruptions and for at least 12 weeks (approximately 5 times the mean terminal t1/2 of luspatercept based on multiple-dose PK data) following IP discontinuation, even if he has undergone a successful vasectomy.

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.] ** Agreement to use highly effective methods of contraception that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly throughout the course of the study. Such methods include: Combined (estrogen and progesterone/progestin containing) hormonal contraception: Oral; Intravaginal; Transdermal; Progestogen/progestin only hormonal contraception associated with inhibition of ovulation: Oral; Injectable hormonal contraception; Implantable hormonal contraception; Placement of an intrauterine device (IUD); Placement of an intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomized partner; Sexual Abstinence.

Exclusion Criteria

* Participant has a diagnosis of Hemoglobin S/β-thalassemia or alpha (α)-thalassemia (eg, Hemoglobin H); β-thalassemia combined with α-thalassemia is allowed.
* Participant has of active hepatitis C (HCV) infection, as demonstrated by a positive HCF-ribonucleic acid (RNS) test of sufficient sensitivity, or active infectious hepatitis B (as demonstrated by the presence of hepatitis B surface antigen (HBsAG) and/or hepatitis B virus (HBV)-deoxyribonucleic acid (DNA) positive, or known positive human immunodeficiency virus (HIV).

Note: Participants receiving antiviral therapies should have 2 negative HCV-RNA tests 3 months apart before ICF/IAF signature, ie, one test at the end of the antiviral therapy and the second test 3 months following the first test.

* Participant has deep vein thrombosis (DVT), stroke, or other thromboembolic event(s) (except clogged indwelling catheter) requiring medical intervention ≤ 24 weeks prior to enrollment.
* Participant has platelet count > 1000 x 109/L.
* Participant has treatment with another investigational drug or device ≤ 28 days prior to enrollment.
* Participant has prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536).
* Participant underwent or is scheduled for HSCT or gene therapy.
* Participant use of iron chelation therapy (ICT), if initiated ≤ 8 weeks prior to enrollment (allowed if initiated > 8 weeks before or during treatment).
* Participant received treatment with hydroxyurea immunomodulatory drugs IMiDs (such as thalidomide), other fetal Hb (HbF) inducers or erythropoiesis-stimulating agents (ESAs) ≤ 12 weeks prior to enrollment for NTD participants and ≤ 24 weeks for TD participants.
* Participant is pregnant or breastfeeding female or plan to get pregnant during the study.
* Participant has uncontrolled hypertension. Controlled hypertension for this protocol is considered: blood pressure value corresponding to ≤ Grade 1 according to NCI CTCAE version 5.0 with or without pharmacological treatment.
* Participant has major organ damage, including:

  1. Symptomatic splenomegaly
  2. Liver disease with alanine aminotransferase (ALT)/aspartate aminotransferase (AST) > 3X the upper limit of normal (ULN) for age
  3. Heart disease, heart failure as classified by the New York Heart Association (NYHA) classification 3 or higher, or significant arrhythmia requiring treatment, or recent myocardial infarction within 6 months of enrollment
  4. Lung disease, including pulmonary fibrosis or pulmonary hypertension of Grade ≥ 3 according to NCI-CTCAE version 5.0.
  5. Renal insufficiency defined as:
* A serum creatinine based on age/gender based on threshold derived from Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control.
* Participant has proteinuria ≥ Grade 3 according to NCI CTCAE version 5.0 (which is equivalent to a urine protein/creatinine ratio > 215 mg/mmol of creatinine), or a urine albumin/creatinine ratio > 129 mg/mmol of creatinine.
* Participant use of high dose long-term therapy with systemic glucocorticoids ≤ 12 weeks prior to enrollment (physiologic replacement therapy for adrenal insufficiency is allowed). Low-dose long-term (defined as ≤ 0.2 mg/kg/day or ≤ 10 mg/day of prednisone equivalent), short treatment (eg, for prevention or treatment of transfusion reactions) inhaled, intranasal and topical corticosteroids are allowed.
* Participant has history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the IP (refer to the IB).
* Participant use of cytotoxic agents, immunosuppressants ≤ 28 days prior to enrollment (ie, antithymocite globulin (ATG) or cyclosporine).
* Participant has history of malignancy with the exception of:

  1. Curatively resected nonmelanoma skin cancer.
  2. Curatively treated carcinoma in situ.
  3. Other solid tumor with no known active disease in the opinion of the Investigator.
* Participant who has extramedullary hematopoiesis (EMH) complications or requires treatment to control the growth of EMH masse(s) during the screening period.
* Participants with any medical or psychiatric condition that in the opinion of the investigator would put the participant at unacceptable risk of participating in the study or may impact interpretation of the study results.
* Participants who use herbs or food supplements (eg: Chinese traditional medicine), if, per investigator's judgment, likely to impact the safety and efficacy assessment, for 24 weeks before initiating the study treatment for TD participants, and 12 weeks for NTD participants.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2035-06-11 (Estimated)

PRIMARY OUTCOMES:
Determination of the Recommended Dose (RD | Cycle 1 up to the day before Cycle 2 Day 1 or Study Day 22 if not receiving the second treatment cycle
  Determine the recommended dose of luspatercept that is safe and tolerable in pediatric participants with transfusion-dependent B-thalassemia or non-transfusion-dependent β-thalassemia
Pharmacokinetics - Cmax | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Maximum serum concentration of drug
Pharmacokinetics - AUC | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Area under the curve
Pharmacokinetics (PK) - t1/2 | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Half-life
Pharmacokinetics (PK) - CL/F | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Apparent oral clearance
Pharmacokinetics (PK) - Vd/F | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Apparent volume of distribution

SECONDARY OUTCOMES:
Mean change in Red Blood Cell (RBC) Transfusion Burden for transfusion-dependent β-thalassemia participants | 12 weeks prior to enrollment; Treatment Period and up to End of Treatment including Long-term Treatment Period - Up to 5 years
  Change from baseline as continuous variable
Mean change in hemoglobin levels for non-transfusion-dependent β-thalassemia participants | 12 weeks prior to enrollment; Treatment Period and up to End of Treatment including Long-term Treatment Period - Up to 5 years
  Change from baseline as continuous variable
Immunogenicity | Time from Cycle 1 Day 1 of Treatment Period up to a maximum of 1 year
  Frequency of antidrug antibodies (ADA)
Mean change from baseline in mean daily dose of iron chelation therapy (ICT) | 12 weeks prior to enrollment; Treatment Period and up to End of Treatment including Long-term Treatment Period - Up to 5 years
  Change from baseline as continuous variable
Mean change from baseline in serum ferritin | 12 weeks prior to enrollment; Treatment Period and up to End of Treatment including Long-term Treatment Period - Up to 5 years
  Change from baseline as continuous variable
Safety - Incidence of Adverse Events (AEs) | From enrollment until at least 9 weeks after last dose of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (2):
  - Local Institution - 601, Los Angeles, California
  - New York Presbyterian Hospital, New York, New York
- China (6):
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - People's Liberation Army The 923rd Hospital, Nanning, GX
  - West China Hospital - Sichuan University, Chengdu, Sichuan
  - Sun Yat-sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Universitatsklinikum Ulm, Ulm
- General Children's Hospital "Agia Sophia", Athens, Greece
- India (6):
  - Kamala Hospital and Research Center, Hyderabad, Andhra Pradesh
  - MCGM - Comprehensive Thalassemia Care, Pediatric Hematology-Oncology & BMT Centre, Borivali (E), Mumbai, Maharashtra
  - Kingsway Hospitals, Nagpur, Maharashtra
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
  - Local Institution - 803, Kolkata
  - Christian Medical College & Hospital, Vellore
- Italy (4):
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, Roma
  - Ente Ospedaliero Ospedali Galliera - Centro della Microcitemia e delle Anemie Congenite, Genoa
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliero Universitaria S. Luigi Gonzaga, Orbassano
- Local Institution - 700, Beirut, Lebanon
- Thailand (3):
  - Chulalongkorn University Faculty of Medicine - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Ramathibodi Hospital, Mahidol University, Phyathai
- Local Institution - 401, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04143724.html